CLINICAL TRIAL: NCT03594539
Title: The Effects of Phosphate on Microvascular Function
Brief Title: Phosphate Microvascular Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: VAH170095
Record Dates: First submitted 2018-07-09; First posted 2018-07-20 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: End Stage Renal Disease; Hyperphosphatemia
Keywords: ESRD; Microvascular; Hyperphosphatemia; LDF
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either lanthanum carbonate or placebo for 2 weeks. They will then be assigned to the other arm of the study. They will be in the alternate arm for 2 weeks and then complete the study,
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacy dispensing the drug will be responsible for generating placebo and distributing drug. The investigators, care providers and patient will not have access to this data. Study outcomes will be comparing arms but not with knowledge of which arm occurred when.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard (No Intervention): Participants will have their hyperphosphatemia managed with lanthanum carbonate 1 g with meals and 500 mg with snacks as per typical care, for 2 weeks.
- Intervention (Placebo Comparator): Participants will take a placebo instead of standard care with a phosphate binder, for 2 weeks.
  Interventions: Other: Withholding standard phosphate binder

INTERVENTIONS:
Other: Withholding standard phosphate binder — In this trial, placebo represents the intervention and not the control. Standard therapy for hyperphosphatemia in end-stage renal disease includes treatment with a phosphate binder. In this trial the intervention will be to withhold the phosphate binder and use placebo instead. In this way the effect of a higher serum phosphate can be evaluated.
  Arms: Intervention

SUMMARY:
Elevated phosphate concentrations in the blood have been associated with multiple negative health outcomes in patients with chronic kidney disease as well as in the general population. These negative outcomes include an increased risk of vascular complications like heart attack and stroke. While complications like heart attack and stroke reflect obstructive disease in large blood vessels, recent evidence suggests that elevated phosphate concentrations may first lead to disease in small blood vessels.

This single site clinical trial will randomize 20 veterans with end stage renal disease on hemodialysis to either a phosphate binder or placebo and evaluated for changes in their microvascular function using laser-Doppler flowmtery and nail-fold capillaroscopy.

DETAILED DESCRIPTION:
Project Background: Recent studies have suggested that increased serum phosphate and phosphate intake may acute impair microvascular blood flow. However, this has never been directly tested using imaging techniques that directly measure microvascular flow. The end-stage renal disease population on hemodialysis at the VA San Diego is an ideal population to evaluate this effect.

Project Question: Does reduction of serum phosphate through the use of a phosphate binder (lanthanum carbonate) increase microvascular blood flow in persons with ESRD? Project Methods: The investigators propose a 4 week, randomized, double-blinded, placebo controlled, single-center, crossover trial. Participants will have their microvascular function assessed at the baseline of the study using laser-Doppler flowmetry and nail-fold capillaroscopy. They will then be randomized to either lanthanum carbonate or placebo for 2 weeks. Microvascular measurements will be repeated at the end of the 2 week period. Participants will then cross-over to the other study arm. After 2 weeks in the other study arm, they will have microvascular measurements repeated and the trial will then be complete. The primary outcome of the study will be the % change in skin blood flow after heating from 31 degrees Celsius to 44 degrees Celsius. This will be compared within each individual after they complete each arm of the study. Changes seen on nail-fold capillaroscopy, acceptability, safety, and adherence will be key secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ESRD on hemodialysis (HD) for >90 days.
* Age >21.
* Capacity to understand and sign informed consent as assess by principal investigator.
* On a phosphate binder with stable dose for >2 weeks.
* Serum phosphate at screening visit of <7.0.

Exclusion Criteria:

* Pregnancy.
* Actively breastfeeding.
* Use of oral contraceptives.
* Inability to take oral medications.
* History of medication non-compliance as assessed by the treating physician.
* Patients currently enrolled in another trial.
* Planned or expected surgical procedure during study period.
* Planned or expected hospitalization during study period.
* Corrected serum calcium greater than 10.2 mg/dl.
* Serum intact PTH >1000 pg/ml
* Albumin < 3 g/dl.
* Allergy or intolerance to lanthanum carbonate.
* Principal investigator deems patient to be unsuitable.
* Non-English speaking persons. (Study performed at VA, therefore do not anticipate this represents a significant portion of the population).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-17 (Estimated)

PRIMARY OUTCOMES:
% Change in flux of blood after skin heating to 44 C as measured using laser-Doppler flowmtery. | Performed at initial study visit, at the end of the first arm of the study (Day 14) and again at the end of the second arm of the study (Day 28)
  Flux of blood through skin will be measured using a Perimed PF5000. This will be performed at baseline in a temperature controlled room. Baseline skin measurements will be made at 31C. Skin will then be heated to 44 C. The percent change will be the outcome. This outcome will be compared within each person at the conclusion of each arm. Measurements will all be made on the Monday or Tuesday, the day of the participant's first dialysis treatment of the week. Measurements will be made prior to dialysis.

SECONDARY OUTCOMES:
Change in capillary count seen post occlusion from pre occlusion, as determined by nail-fold capillaroscopy. | Performed at initial study visit, at the end of the first arm of the study (Day 14) and again at the end of the second arm of the study (Day 28)
  Participants will undergo nail fold capillaroscopy using a CapiScope (KK Technology, Honiton United Kingdom) at baseline and then at the end of each treatment arm. Using a capillarascope a capillary count will be made. After measurement a BP cuff will be inflated to 200 mm Hg occlude flow to a single digit for 1 minute. 30 sec after release the count will be made again. This change will be compared within individuals between measurements made at the completion of each arm in the study. Measurements will all be made on the Monday or Tuesday, the day of the participant's first dialysis treatment of the week. Measurements will be made prior to dialysis. Values at the end of each treatment arm will be compared.

IPD SHARING:
Plan to Share IPD: Yes
de-identified data may be shared at end of study
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] O'Seaghdha CM, Hwang SJ, Muntner P, Melamed ML, Fox CS. Serum phosphorus predicts incident chronic kidney disease and end-stage renal disease. Nephrol Dial Transplant. 2011 Sep;26(9):2885-90. doi: 10.1093/ndt/gfq808. Epub 2011 Feb 3. PMID 21292817
- [Background] Thambyrajah J, Landray MJ, McGlynn FJ, Jones HJ, Wheeler DC, Townend JN. Abnormalities of endothelial function in patients with predialysis renal failure. Heart. 2000 Feb;83(2):205-9. doi: 10.1136/heart.83.2.205. PMID 10648498
- [Background] Stevens KK, Denby L, Patel RK, Mark PB, Kettlewell S, Smith GL, Clancy MJ, Delles C, Jardine AG. Deleterious effects of phosphate on vascular and endothelial function via disruption to the nitric oxide pathway. Nephrol Dial Transplant. 2017 Oct 1;32(10):1617-1627. doi: 10.1093/ndt/gfw252. PMID 27448672